CLINICAL TRIAL: NCT05805774
Title: pDIFFIR: Geriatric Periprosthetic DIstal Femur: FIxation Versus Replacement - A Randomized Controlled Trial of Acute Open Reduction Internal Fixation (ORIF) Versus Distal Femur Replacement (DFR)
Brief Title: pDIFFIR: Geriatric Periprosthetic DIstal Femur: FIxation Versus Replacement
Acronym: pDIFFIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-001
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Distal Femur Fracture; Periprosthetic Fracture Around Prosthetic Joint Implant Knee; Knee Fracture
Keywords: Periprosthetic Distal Femur fracture; Knee replacement; Surgical fixation; Geriatric patients
MeSH Terms: conditions — Femoral Fractures, Distal; Knee Fractures | interventions — Surgical Fixation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - DFR (Active Comparator)
  Interventions: Procedure: Distal Femur Replacement
- Group B - ORIF (Active Comparator)
  Interventions: Procedure: Surgical fixation

INTERVENTIONS:
Procedure: Distal Femur Replacement — Knee surgery to remove the lower part of the femur and knee joint (where the broken bones are) and will replace them with an artificial knee joint (prosthesis).
  Arms: Group A - DFR
Procedure: Surgical fixation — Knee surgery to fix the fracture, that can use wires, nails, screws, pins or plates to health and fix the bones together.
  Arms: Group B - ORIF

SUMMARY:
Periprosthetic distal femur fractures are a significant source of morbidity and mortality for elderly patients. One treatment option involved a surgical fixation with plates or nails, screws and cables/wires along the side of your fractured bone. The second method consists in replacing your knee joint with an artificial knee prosthesis (artificial knee joint).

The primary objective is to determine if acute distal femur replacement improves knee pain and functional outcomes compared to surgical fixation. Secondary outcomes are mortality, reoperation, complications, post-operative pain and quality of life. A health economic analysis will be conducted to assess the cost-effectiveness of both treatments.

A total of 148 patients (74/group) will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* • 65 years and older

  * Isolated periprosthetic fracture of the distal femur around a stable primary total knee arthroplasty (Lewis and Rorabeck Type 1-2)
  * Fracture is acute (within 1 week from time of injury)
  * Patient was ambulatory (with or without walking aids) in the community and at home prior to the injury
  * Independent or moderately frail with score of 3 to 6 on the validated Clinical Frailty Scale
  * Patient is able to read and understand the consent form document, or an interpreter is available to the patient at the time of consent and follow-up
  * Patient or substitute decision maker is able to provide written informed consent to participate in the study

Exclusion Criteria:

* • Active infection around the fracture (soft tissue or bone)

  * Open fracture
  * Bilateral femur fractures
  * Major neuro-vascular injury requiring intervention, compartment syndrome and major neurologic injuries
  * Pathological fracture excluding osteoporosis
  * Ipsilateral total knee arthroplasty using revision components (varus/valgus constraint, stemmed femoral components)
  * Periprosthetic distal femur fracture around a loose or failing primary total knee arthroplasty (Lewis and Rorabeck Type III)
  * Ipsilateral primary partial knee or patellofemoral arthroplasty
  * Previous ORIF of the distal femur or proximal tibia or patella
  * Current or previous extensor mechanism (patellar tendon, quadriceps tendon, or patella fracture) disruption or repair
  * Poly-trauma status (Injury Severity Score>15) or any associated major injuries of the lower extremities that may hinder post-operative ambulation
  * Medical contraindication to surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2030-12-10 (Estimated); Study Completion 2032-12-10 (Estimated)

PRIMARY OUTCOMES:
Knee function | 12 months
  Compare knee pain between the two groups using the Oxford Knee Score - which is a patient reported outcome measure. It assess knee function and gives a rating from 0 to 48 - being 0 bad knee function and 48 - excellent knee function.

SECONDARY OUTCOMES:
Mortality | 24 months
  Track patient's death.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Khoshbin, MD, Principal Investigator — Unity Health Toronto - St Michael's Hospital; Jesse Wolfstadt, MD, Principal Investigator — Mount Sinai Health Hospital
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided